CLINICAL TRIAL: NCT01297946
Title: An Open-label, Randomized, Two-way, Cross-over Study to Assess the Efficacy of Dual-hormone Closed-loop Strategy as Compared to Conventional CSII Therapy in Regulating Glucose Levels in Adults With Type-1 Diabetes in the Context of Exercise
Brief Title: Closed-loop Control of Glucose Levels in the Context of Exercise in Adults With Type-1 Diabetes
Acronym: CLASS-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: McGill University (Other); Montreal Children's Hospital of the MUHC (Other); Diabetes Québec (Other); Medtronic Minimed (Unknown)
Responsible Party: Rémi Rabasa-Lhoret, M.D., Ph.D., Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-01
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open-loop (Placebo Comparator): Conventional continuous subcutaneous insulin infusion (CSII) therapy
  Interventions: Device: Conventional continuous subcutaneous insulin infusion therapy
- Dual-hormone closed-loop (Experimental): Variable subcutaneous insulin and glucagon infusion rates will be used to regulate glucose levels. The infusion rates are based on continuous glucose sensor reading and a control algorithm.
  Interventions: Device: Dual-hormone closed-loop

INTERVENTIONS:
Device: Conventional continuous subcutaneous insulin infusion therapy
  Arms: Open-loop
Device: Dual-hormone closed-loop
  Arms: Dual-hormone closed-loop

SUMMARY:
Recent developments of continuous glucose sensors and insulin infusion pumps have motivated the research toward closed-loop strategies to regulate glucose levels in patients with type 1 diabetes. In a closed-loop strategy, the pump(s) infusion rate is altered based on a computer-generated recommendation that relies on continuous glucose sensor readings. In this study, we aim to compare the effectiveness of dual-hormone (insulin+glucagon) closed-loop strategy to open-loop conventional continuous subcutaneous insulin infusion pump (CSII) therapy in regulating glucose levels during an evening exercise and on a night following an exercise in adults with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for at least one year.
* On insulin pump therapy for at least 3 months.
* HbA1c ≤ 10%.

Exclusion Criteria:

* Clinically significant nephropathy, neuropathy or retinopathy.
* Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* A recent injury to body or limb, muscular disorder, use of any medication or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the exercise protocol.
* Pregnancy.
* Severe hypoglycemic episode within two weeks of screening.
* Current use of glucocorticoid medication (by any route of administration except low dose stable inhaled).
* Known or suspected allergy to the trial products or meal contents.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
* Anticipating a significant change in exercise regimen between admissions (i.e. starting or stopping an organized sport).
* Failure to comply with team's recommendations (e.g. not willing to eat snack, not willing to change pump parameters, etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)

PRIMARY OUTCOMES:
Percentage of time of plasma glucose concentrations spent in target range (4.0-10.0 mmol/l from 4:00p.m.-11:00p.m. and 4.0-8.0 mmol/l from 11:00p.m.-7:00a.m.) | 4 p.m. - 7 a.m.

SECONDARY OUTCOMES:
Percentage of time of plasma glucose concentrations spent in the low range (< 4.0 mmol/l). | 4 p.m. - 7 a.m.
Percentage of time of plasma glucose concentrations spent in the high range (>10.0 mmol/l from 4:00p.m.-11:00 p.m. and >8.0 mmol/l from 11:00 p.m.-7:00 a.m.). | 4 p.m. - 7 a.m
Percentage of overnight time of plasma glucose concentrations spent in target range (4.0 - 8.0 mmol/l). | 11 p.m. - 7 a.m.
Percentage of overnight time of plasma glucose concentrations spent in the low range ( < 4.0 mmol/l). | 11 p.m. - 7 a.m.
Percentage of overnight time of plasma glucose concentrations spent in the high range (above 8 mmol/l). | 11 p.m. - 7 a.m.
Total insulin delivery. | 4 p.m. - 7 a.m.
Total overnight insulin delivery (11 p.m. - 7 a.m.). | 11 p.m. - 7 a.m.
Standard deviation and/or MAGE (Mean Amplitude of Glycemic Excursions) index of plasma glucose concentrations as measures of glucose variability. | 4 p.m. - 7 a.m.
Number of subjects with at least one plasma glucose measurement less than 3.9 mmol/l. | 4 p.m. - 7 a.m.
Number of subjects with at least one overnight plasma glucose measurement less than 3.9 mmol/l. | 11 p.m. - 7 a.m
Number of subjects with at least one exercise-induced plasma glucose measurement less than 3.9 mmol/l. | 5:50 p.m. - 7:20 p.m
Number of subjects with as at least one plasma glucose measurement below 3.3 mmol/l. | 4 p.m. - 7 a.m.
Number of subjects with at least one overnight plasma glucose measurement below 3.3 mmol/l. | 11 p.m. - 7 a.m
Number of subjects with at least one exercise-induced plasma glucose measurement below 3.3 mmol/l. | 5:50 p.m. - 7:20 p.m
Number of subjects with as at least one plasma glucose measurement below 3.0 mmol/l. | 4 p.m. - 7 a.m.
Number of subjects with at least one overnight plasma glucose measurement below 3.0 mmol/l. | 11 p.m. - 7 a.m
Number of subjects with at least one exercise-induced plasma glucose measurement below 3.0 mmol/l. | 5:50 p.m. - 7:20 p.m

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, M.D., Ph.D., Principal Investigator — Institut de Recherches Cliniques de Montréal (IRCM)
Locations (1):
- Institut de Recherches Cliniques de Montréal (IRCM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Heyland DK, Heyland R, Bailey A, Howard M. A novel decision aid to help plan for serious illness: a multisite randomized trial. CMAJ Open. 2020 Apr 28;8(2):E289-E296. doi: 10.9778/cmajo.20190179. Print 2020 Apr-Jun. PMID 32345707
- [Derived] Haidar A, Legault L, Dallaire M, Alkhateeb A, Coriati A, Messier V, Cheng P, Millette M, Boulet B, Rabasa-Lhoret R. Glucose-responsive insulin and glucagon delivery (dual-hormone artificial pancreas) in adults with type 1 diabetes: a randomized crossover controlled trial. CMAJ. 2013 Mar 5;185(4):297-305. doi: 10.1503/cmaj.121265. Epub 2013 Jan 28. PMID 23359039